CLINICAL TRIAL: NCT00985569
Title: Surveying The Outcomes Of Lubiprostone (The STOOL Study): The Effect of Lubiprostone on Reducing the Number of Medications Prescribed to Nursing Home Residents and Its Impact on Selected Quality Indicators
Brief Title: Surveying The Outcomes Of Lubiprostone (The STOOL Study) in Nursing Home Residents
Acronym: STOOL
Status: Withdrawn | Type: Observational
Why Stopped: Enrollment was never begun.
Sponsor: Synergy Health Solutions (Other)
Responsible Party: Malcolm Fraser, MD, CMD, Synergy Health Solutions
Other Study IDs: STOOL
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Constipation
Keywords: Constipation; Nursing Home; Quality Indicator
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lubiprostone: Subjects switching from current bowel medicines to lubiprostone

SUMMARY:
The purpose is to assess the efficacy, clinical outcomes, and potential Quality Indicator benefits associated with the use of Lubiprostone in nursing home residents with a confirmed diagnosis of chronic idiopathic constipation.

DETAILED DESCRIPTION:
The study is a prospective, observational, open-label, non-placebo, controlled study to measure the effects of Lubiprostone on CIC in nursing home residents. All clinical sites will follow a common protocol using standardizes definitions in which eligible patients will be asked to participate in the proposed study. During the course of the study, various selected parameters will be measured and compared to establish the clinical efficacy of Lubiprostone in the treatment of CIC.

The study sample (N=105) will be comprised of nursing home residents with a confirmed diagnosis of CIC. A power analysis generated a sample size of 97 residents. To protect the validity of the test, 8 residents were added to the final study sample to allow for losses to followup. Therefore, a final sample size of 105 residents was identified for the study.

Patients meeting the inclusion criteria will be recruited for participation in the study. 3 sites in Central Florida with multiple Nursing Homes per site will be recruited to participate in the proposed study.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for the study:

* Adult men and women nursing home residents;
* Confirmed diagnosis of CIC using Rome criteria;
* Prescribed two or more laxatives, at recruitment;
* Taking 9 or more oral medicines (including prescription, OTC and prn)
* Free from conditions likely to be fatal within six months;
* Able to read or understand English; and
* Able and willing to provide informed consent or has a guardian/agent who can provide consent.

Exclusion Criteria:

* Currently pregnant;
* Presence of megacolon;
* Presence of rectal sigmoid cancer;
* Presence of colon cancer;
* Presence of anal incompetence;
* Conditions likely to be fatal within six months;
* Taking 8 or fewer medicines;
* Enrolled in hospice;
* Non-English speaking patients; and
* Unwilling or unable to provide informed consent and has no guardian/agent.
* Expected to be discharged within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nursing Home Residents (adult subjects living in Nursing Homes)
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-04 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
To determine the overall reduction in the number of oral medicines taken by each NH resident at enrollment and at 60 days. | 60 days

SECONDARY OUTCOMES:
Reduce the number of oral medicines being taken by any nursing home resident from 9 or more to fewer than 9. (Quality Indicator Number 6) | 60 days
To compare the occurrence of fecal impaction during a 60-day period prior to initiating Lubiprostone with a 60 day period after initiating Lubiprostone. (Quality Indicator Number 11) | 60 days
To compare the occurrence of fecal incontinence during a 60-day period prior to initiating Lubiprostone with a 60 day period after initiating Lubiprostone. | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm R Fraser, MD, Principal Investigator — Synergy Health Solutions
Locations (3):
- United States (3):
  - Geriatric Medical Associates, Brooksville, Florida
  - Cassellberry Family Practice, Casselberry, Florida
  - Osler Geriatrics, Melbourne, Florida